CLINICAL TRIAL: NCT03215043
Title: Evaluation of Metabolic Parameters in Subjects With Intermediate Hyperglycemia Supplemented With Eriocitrin: A Parallel, Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Effect of Eriocitrin Supplementation in Subjects With Intermediate Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thais Cesar (Other)
Collaborators: Ingredients by Nature TM (Unknown)
Responsible Party: Sponsor-Investigator, Thais Cesar, Principal Investigator, São Paulo State University
Organization: São Paulo State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SaoPSU7
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pre Diabetes
Keywords: Eriocitrin; Intermediate hyperglycemia; Citrus bioflavonoids
MeSH Terms: conditions — Glucose Intolerance | interventions — eriocitrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Individuals will receive a dose of 140 mg / d eriocitrin for 12 weeks
  Interventions: Dietary Supplement: Eriocitrin
- Group B (Experimental): Individuals will receive a dose of 280 mg / d eriocitrin for 12 weeks
  Interventions: Dietary Supplement: Eriocitrin
- Group C (Experimental): Individuals will receive a dose of 560 mg / d eriocitrin for 12 weeks
  Interventions: Dietary Supplement: Eriocitrin
- Group D (Placebo Comparator): Individuals will receive the placebo with corn starch excipient for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Eriocitrin — The selected individuals will be randomly distributed in 4 groups through random number generator program. Group A (n = 20) will receive a dose of 140 mg / d eriocitrin; Group B (n = 20) eriocitrin 280 mg / d; The C group (n = 20) 560 mg / d eriocitrin; And group D (n = 20) will receive the placebo with corn starch excipient. All doses will be packaged in Manipulation Pharmacy, and should be of the same type, color and size. Individuals will be instructed to regularly ingest a pre-dinner capsule for 12 weeks.
  Arms: Group A; Group B; Group C
Other: Placebo — The selected individuals will be randomly distributed in 4 groups through random number generator program. Group A (n = 20) will receive a dose of 140 mg / d eriocitrin; Group B (n = 20) eriocitrin 280 mg / d; The C group (n = 20) 560 mg / d eriocitrin; And group D (n = 20) will receive the placebo with corn starch excipient. All doses will be packaged in Manipulation Pharmacy, and should be of the same type, color and size. Individuals will be instructed to regularly ingest a pre-dinner capsule for 12 weeks.
  Arms: Group D

SUMMARY:
First, it will be evaluated whether supplementation of eriocitrin reduces hyperglycemia and insulin resistance, significantly reducing the risk of diabetes. The effects of eriocitrin on the lipid profile, inflammatory, endothelial, hepatic and renal biomarkers will also be evaluated. It is expected that metabolic parameters that constitute risk factors for diabetes and associated chronic diseases are expected to be improved by supplementation with eriocitrin

DETAILED DESCRIPTION:
Volunteers will be invited to appear in a 12-hour fast to measure glucose levels, glycated hemoglobin and to perform the glucose tolerance test, in addition to an individual interview to confirm eligibility according to the inclusion and exclusion criteria. The collection of blood and the glycemic curves will be carried out next to a Laboratory of Clinical Analyzes, commercial, based in the city of Araraquara.

The sample number took into account variances on glycated hemoglobin with a type I error α = 0.05 and a type II error β = 0.2 (80% power) (Mohammad, 2015). The minimum sample size considering an approximately 20% dropout rate, should have 20 individuals per group.

In order to ensure adequate nutrition for the nutritional and energetic needs of volunteers, an individual food plan shall be prescribed, calculated according to the DRI equations. The volunteer will be asked to complete the Food Record for three days at the 3rd, 5th, 7th, 9th and 11th week. Data analysis of energy intake, macronutrients and micronutrients will be performed through the DietBox® . The anthropometric measurements will be performed before the intervention and in the 3rd, 5th, 7th, 9th and 11th week by Nutritionist. Four samples of 30mL of fasting blood each will be obtained before the intervention, in the 4th, 8th and 12th week in the Laboratory of Clinical Analyzes. The blood will be centrifuged to obtain the serum, which will be frozen at -80 ° C until subsequent biochemical analyzes.

Normality and homogeneity will be evaluated by Shapiro-Wilk test and Levine tests, respectively. The T test will be used to compare baseline time between groups. The two-way repeated-measures ANOVA will be used to compare changes within and between the eriocitrin and control groups over the 12-week period. P significant at ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Glycemia of 6.1 to 7.0 mmol / L
* Glycated hemoglobin with values between 5.7 and 6.4%

Exclusion Criteria:

* use of drugs, vitamins and dietary supplements, alcohol consumption (> 20 g alcohol/d), and intense physical activity (> 5 hours/week).
* History of cardiovascular disease, diabetes mellitus, liver or kidney disease

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Glucose | 12 Weeks
  mg/dL

SECONDARY OUTCOMES:
glycated hemoglobin | 12 Weeks
  percentage
insulin | 12 Weeks
  µU/mL
Cholesterol | 12 Weeks
  mg/dL
triglycerides | 12 Weeks
  mg/dL
HDL-C | 12 Weeks
  mg/dL
LDL-C | 12 Weeks
  mg/dL
TNF-alpha | 12 Weeks
  pg.mL
Interleucina 6 | 12 Weeks
  pg.mL
c-reactive protein | 12 Weeks
  mg/dL
aspartate aminotransferase | 12 Weeks
  U/L
alkaline phosphatase | 12 Weeks
  U/L
Gamma-Glutamyl Transferase | 12 Weeks
  U/L
alanine aminotransferase | 12 Weeks
  U/L

OTHER OUTCOMES:
Body mass | 12 Weeks
  Kg
fat mass | 12 Weeks
  kg
percentage of total body fat | 12 Weeks
  Percentage
visceral fat area | 12 Weeks
  cm2

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, Ph.D, Principal Investigator — Sao Paulo State University "Julio de Mesquita Filho", Faculdade de Ciências Farmacêuticas
Locations (1):
- Sao Paulo State University "Julio de Mesquita Filho", Faculdade de Ciências Farmacêuticas, Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
There is still no decision regarding if the individual participant data (IPD) will be available to other researchers.

REFERENCES:
- [Background] Mohammad M, et al. Effects of Hesperidin Supplementation on Glycemic Control, Lipid Profile and Inflammatory Markers in Patients with Type 2 Diabetes: A Randomized Double Blind Placebo Control Clinical Trial. Research Article, Acta Biologica Indica 2015, 4(1):75-83. ISSN 2279-0160
- See also: WHO, 2006 - Definition and diagnosis of diabetes mellitus and intermediate hyperglycemia. — https://www.who.int/publications/i/item/definition-and-diagnosis-of-diabetes-mellitus-and-intermediate-hyperglycaemia